CLINICAL TRIAL: NCT04938310
Title: Impact of Wearing a Support Garment on Mobility, Functional Capacity, Self-esteem, Quality of Life and Skin Maceration Following Parietal Gastrectomy
Brief Title: Impact of Wearing a Support Garment Following Parietal Gastrectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped prematurely by sponsor due to lack of funding following company closure
Sponsor: Laval University (Other)
Collaborators: Bodynov (Unknown); Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Laurent Biertho, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bodynov
Record Dates: First submitted 2021-05-28; First posted 2021-06-24 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Obesity, Morbid
Keywords: Bariatric surgery
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Sleeve gastrectomy
  Interventions: Procedure: sleeve gastrectomy
- Support garment group (Experimental): Sleeve gastrectomy followed by a period of 12-month with a support garment
  Interventions: Procedure: sleeve gastrectomy; Device: support garment

INTERVENTIONS:
Procedure: sleeve gastrectomy — sleeve gastrectomy
Device: support garment — A custom made support garment
  Arms: Support garment group

SUMMARY:
Custom-made orthopedic support equipment and abdominal-lumbar support belts offer promising potential for several aspects affecting the health and well-being of people with obesity who choose a surgical weight loss option. However, research is needed to quantitatively document their short and long term effects on a wide range of parameters related to mobility, quality of life, lower back pain and skin maceration following parietal gastrectomy. The objective of this study is to characterize the effect of a support garment in an experimental design where a subgroup of participants will be randomized and followed for the first 12 months after a gastrectomy. The measures will be: physical activity, lower back pain, self-esteem, quality of life, skin maceration and infections. This study will scientifically document the usefulness and effectiveness of support garments throughout the weight loss surgery process.

ELIGIBILITY:
Inclusion Criteria:

* meeting the NIH criteria for bariatric surgery
* BMI >= 35 kg/m2

Exclusion Criteria:

* chronic pulmonary obstructive disease
* gastric stoma
* psychiatric disease contraindicated for bariatric surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Excess skin | From baseline to 12 month following sleeve gastrectomy
  Excess skin measured with the Iglesias scale, scores are from 1 to 5, higher score means a worse excess skin
Skin maceration | From baseline to 12 month following sleeve gastrectomy
  maceration evaluated with an in-house questionnaire reported as presence or absence of skin maceration
Skin infection | From baseline to 12 month following sleeve gastrectomy
  infection evaluated with an in-house questionnaire reported as presence or absence of skin infection
Impact of excess skin | From baseline to 12 month following sleeve gastrectomy
  Sahlgrenska Excess Skin questionnaire assesses excess skin after weight loss for specific body parts and body as a hole. Inconvenience of excess skin is evaluated on a scale from 0 to 10, higher score means higher perception that the excess skin is an inconvenience.
Physical activity | From baseline to 12 month following sleeve gastrectomy
  Physical activity evaluated by wearing an activity monitor
Physical activity | From baseline to 12 month following sleeve gastrectomy
  Global Physical Activity Questionnaire
Lower back pain | From baseline to 12 month following sleeve gastrectomy
  Quebec back pain scale, scores are from 0 to 100, higher score means greater difficulty in carrying out activities due to low back pain
Self esteem | From baseline to 12 month following sleeve gastrectomy
  Rosenberg self esteem scale, scores are from 10 to 40, higher score mean a stronger self esteem
Self esteem related to physical appearance | From baseline to 12 month following sleeve gastrectomy
  Body Esteem Scale for Adolescent and Adults contains 3 subscales for weight, appearance and attribution. Scores are from 1 to 5, higher score means higher self esteem.
Body image | From baseline to 12 month following sleeve gastrectomy
  Gender-specific body-size guide is a pictorial method of assessing the perception of weight status. It consists of 10 standardized images of adults with known BMI values and is a validated body size perception tool. The scale is gender specific and images range from underweight (BMI <18.5) to class III obesity (BMI> = 40) with approximately a 3 point difference in BMI between the figures on the scale.
Body image | From baseline to 12 month following sleeve gastrectomy
  body shape questionnaire, scores are from 34 to 204, higher score means worse feeling about the appearance.
Body image | From baseline to 12 month following sleeve gastrectomy
  Eating Disorders Examination Questionnaire contains subscales for restraint, eating concern, shape concern and weight concern. Each subscales and global scale scores are form 0 to 6, higher score means worse outcome
Severity of depression symptoms | From baseline to 12 month following sleeve gastrectomy
  Beck Depression Inventory II questionnaire, scores are from 0 to 63, higher score means more severe depressive symptoms.
Anxiety | From baseline to 12 month following sleeve gastrectomy
  State-Trait Anxiety Inventory contains 2 subscales for usual emotional state and current emotional state. Scores are from 20 to 80, higher scores means higher anxiety state.
Social Physique Anxiety | From baseline to 12 month following sleeve gastrectomy
  Social Physique Anxiety Scale, scores are from 12 to 60, higher score means more anxiety
Quality of life | From baseline to 12 month following sleeve gastrectomy
  Laval questionnaire contains 6 subscales for symptoms, activity/mobility, personal hygiene/clothing, emotions, social interactions, and sex life. scores are from 1 to 7, higher score means higher quality of life in each domain
marital satisfaction | From baseline to 12 month following sleeve gastrectomy
  Dyadic adjustment scale, scores are from 0 to 151, higher score indicates a higher level of marital functioning
social ideals of physical appearance | From baseline to 12 month following sleeve gastrectomy
  Sociocultural Attitude Towards Appearance Questionnaire-4 contains 6 subscales (internalization: thinness / low fat mass, internalization: muscular, internalization: general attractiveness, pressures: family, pressures: media, pressures: similar and other significant). Scores are from 1 to 5, higher scores indicating greater internalization and endorsement of societal appearance ideals
gastroesophageal reflux disease | From baseline to 12 month following sleeve gastrectomy
  GastroEsophageal Reflux Disease Score, scores are from 0 to 96, higher score indicates worse gastroesophageal reflux symptoms
adherence in wearing the support garment | From baseline to 12 month following sleeve gastrectomy
  adherence in wearing the support garment evaluated with an adherence journal. Adherence will be calculated as a percentage from the total number of days the participant wears the garment out of the total for the intervention.
persistence in wearing the support garment | From baseline to 12 month following sleeve gastrectomy
  persistence in wearing the support garment will be calculated as a percentage by reporting the number of participants who have stopped wearing the garment compared to those who have used it.
Body composition | From baseline to 12 month following sleeve gastrectomy
  body fat composition assessed by impedance

CONTACTS AND LOCATIONS:
Locations (1):
- Criucpq-Ul, Québec, Quebec, Canada